CLINICAL TRIAL: NCT05299684
Title: The Effect of Smartphone Addiction on the Musculoskeletal System
Brief Title: Smartphone Addiction and Muscular Disorder
Status: Completed | Type: Observational
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Özden Laçin, lecturer, Istanbul Arel University
Other Study IDs: smartphoneaddictionozden
Record Dates: First submitted 2022-03-08; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Myofascial Trigger Point
Keywords: Smartphone; mobile phone addiction; myofascial trigger point; forward head
MeSH Terms: conditions — Technology Addiction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EVALUATION — The level of addiction was assessed with the Smartphone Addiction Scale Short Form (SAS-SF). The posture of participants was evaluated by New York Posture Rating Chart (NYPRC), mostly usage smartphone posture, forward head and myofascial trigger points were questioned according to Simon and Travel criteria. Mann-Whitney U test Pearson's chi-squared test were used for analyzing the data.

SUMMARY:
Background and aim: The use of smartphones, which has reached the level of addiction causes some physical and psychological health problems. The aim was to examine the musculoskeletal disorders of the neck and upper extremities of mobile phone addiction in a population of young adults.

Methods: The study is a cross sectional research conducted on students of a university in İstanbul between December 2018-October 2020. The level of addiction was assessed with the Smartphone Addiction Scale Short Form (SAS-SF). The posture of participants was evaluated by New York Posture Rating Chart (NYPRC), mostly usage smartphone posture, forward head and myofascial trigger points were questioned according to Simon and Travel criteria. Mann-Whitney U test Pearson's chi-squared test were used for analyzing the data.

ELIGIBILITY:
Inclusion Criteria:

* used smartphones
* volunteered to participate in the study.

Exclusion Criteria:

* having any history of trauma at the neck region within the last six months,
* taking any treatment for trigger points within the last 3 months
* having a history of neck surgery.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants of this study included 136 healthy students between the ages of 18 - 25 years. The study group consisted of 84 females and 52 males.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Smartphone Addiction | Baseline
  Smartphone Addictive Scale - Short Form (SAS - SF) that developed by Kwan et al. (2013), was used for the assessment of smartphone addiction. The cut off value of SAS-SF are 31 for men, 33 for women (6). The Turkish translated version of the SAS - SF is a reliable, consistent and valid instrument
Posture | Baseline
  The posture of the participants was assessed by using the New York Posture Rating Chart (NYPRC). In this evaluation method, postural changes that may occur in 13 different parts of the body (head, neck, shoulder, scapula, upper thoracic, waist, rips, abdomen, hips, knees, legs, feet and toe) are observed and scored. Each body segment was scored on the scale of; 5 (correct posture), 3 (slight deviation), or 1 (pronounced deviation). Higher points show better postural alignment
myofascial trigger point | Baseline
  The presence of myofascial trigger points were questioned by Simon and Travel's criteria in the sternocleidomastoid, upper trapezius, levator scapula, rhomboid, infraspinatus and cervical extensor muscles. These criteria were -The presence of a tender spot in a taut band or nodules of skeletal muscle; -Subject recognition of pain upon palpation of a tender spot; -Subject referred pain pattern; -The presence of a local twitch response
Forward head posture | Baseline
  Forward head postures of the participants were evaluated by measuring the tragus to wall distance with a tape measure. For forward head posture, the patients were measured in standing position, leaning against the back wall, in free posture

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Arel University, Istanbul, Turkey (Türkiye)